CLINICAL TRIAL: NCT00628030
Title: Parent Skills Training to Enhance Weight Loss in Overweight Children
Brief Title: NOURISH: Nourishing Our Understanding of Role Modeling to Improve Support and Health
Acronym: NOURISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PT101376; 1R03HD056050-01A1 (NIH)
Record Dates: First submitted 2008-02-22; First posted 2008-03-04 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Pediatric Obesity
Keywords: Behavioral intervention; Obesity prevention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NOURISH (Experimental): The first 2 waves and second 2 waves of participants will receive a 12 and 6 week face-to-face intervention (NOURISH), respectively. The interventions differ only in duration. They cover the same concepts which are grounded in Social Cognitive Theory (SCT). Throughout the interventions the influence of social learning on behavioral outcomes (e.g., parent's modeling of healthy behavior) will be emphasized. Weekly topics provide information about implementing healthy lifestyle behaviors, authoritarian parenting approaches, and strategies for overcoming barriers to change. Parents will receive pedometers for themselves and 1 of their children. A one-hour booster session will be available for all intervention participants 2 months after completion of the interventions.
  Interventions: Behavioral: NOURISH
- Wellness Group (Placebo Comparator): The placebo control group will attend a group session moderated by an independent interventionist. This interventionist will be blinded to the Specific Aims and hypotheses of this study. The session will address the role of diet and exercise in pediatric overweight. In addition, control parents will receive pedometers (and instructions on their use) for themselves and 1 of their children. Finally, control participants will be mailed publicly available brochures on pediatric overweight on 2 occasions during the study. Control participants will also be sent home one additional packet of information (essentially a review of previous mail outs) 2 months after post-testing.
  Interventions: Other: Wellness Group

INTERVENTIONS:
Behavioral: NOURISH — Participants in the NOURISH intervention will have 6 weekly face-to-face parent group sessions regarding healthy eating and physical activity.
  Arms: NOURISH
Other: Wellness Group — Participants in the Wellness Group will have one face-to-face group meeting and information regarding healthy eating and physical activity will be provided on a regular basis via mail.
  Arms: Wellness Group

SUMMARY:
The percentage of overweight children between the ages of 6 and 11 has nearly tripled in the last three decades, and rates are even higher among African Americans.Overweight children are at-risk for numerous health problems, thus effective treatments are urgently needed. This study will evaluate an innovative intervention for ethnically diverse parents (NOURISH), which focuses on helping parents role model and teach their children healthy behaviors.

DETAILED DESCRIPTION:
Pediatric overweight is a national public health concern. The percentage of overweight children in the U.S. between the ages of 6 and 11 has nearly tripled in the last 3 decades. African American children are particularly at risk. Pediatric overweight is associated with numerous physical and psychological health problems. Moreover, overweight children are at significant risk for obesity in adulthood. Thus, a focus on pediatric overweight is an important step in the prevention of adult obesity.

Despite the urgent need for pediatric overweight interventions, outcomes of some of the most rigorous treatments are, at best, mixed. Although research has found that including parents in interventions for pediatric overweight has positive effects on outcomes, parental involvement is usually limited. Moreover, relatively few studies have included sufficient numbers of lower-SES, African American participants, a group at increased risk for pediatric overweight and associated complications. This study will evaluate the efficacy of an intensive intervention targeting ethnically diverse parents of overweight, children ages 6-11 (NOURISH-Nourishing Our Understanding of Role Modeling to Improve Support and Health).

ELIGIBILITY:
Inclusion Criteria:

* To qualify for participation, parents/caregivers must have a child between the ages of 6 and 11 with a BMI > the 85th percentile [128].
* This child must also primarily reside in the participating caregiver's home.
* Participants also need to speak English fluently, and be able to understand and follow basic instructions and perform simple exercises.

Exclusion Criteria:

* Caregivers are ineligible if they are:

  1. non-ambulatory,
  2. pregnant,
  3. or have a clinical diagnosis that may be negatively impacted by exercise.
* Parents whose children have a medical condition or developmental disorder that precludes weight loss using conventional diet and exercise methods are also ineligible for participation.

All parents meeting study criteria will be offered participation in the randomized trial comparing NOURISH with a control group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne E. Mazzeo, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NOURISH: Only parents participated in the weekly intervention. Intervention content was grounded in Social Cognitive Theory (SCT); the influence of social learning on behavioral outcomes (e.g., parent's modeling of healthy behavior) was emphasized. Weekly topics included implementing healthy lifestyle behaviors, authoritarian parenting approaches, and strategies for overcoming barriers to change. Parents received pedometers for themselves and 1 of their children. The first 2 waves and second 2 waves of participants received a 12 and 6 week face-to-face intervention (NOURISH), respectively. A one-hour booster session was available for all intervention participants 2 months after completion of the interventions.
- Wellness Group: Only parents participated in the placebo control group which involved attending a group session moderated by an independent interventionist. This interventionist was blinded to the Specific Aims and hypotheses of this study. The session addressed the role of diet and exercise in pediatric overweight. In addition, control parents received pedometers (and instructions on their use) for themselves and 1 of their children. Finally, control participants were mailed publicly available brochures on pediatric overweight on 2 occasions during the study. Control participants were also sent one additional packet of information (essentially a review of previous mail outs) 2 months after post-testing.
Period: Baseline to Post-Assessment
Arm/Group | NOURISH | Wellness Group
Started | 92 | 92
Completed | 59 | 63
Not Completed | 33 | 29
Not completed — Lost to Follow-up | 28 | 29
Not completed — Withdrawal by Subject | 5 | 0
Period: Post to 6 Month Follow-up
Arm/Group | NOURISH | Wellness Group
Started | 59 | 63
Completed | 27 | 33
Not Completed | 32 | 30
Not completed — Lost to Follow-up | 32 | 30

BASELINE CHARACTERISTICS:
Population: Families completed baseline, post, and six-month follow-up assessments. Although baseline and outcome data for parents and children were collected, only parents participated in the intervention: NOURISH (n = 92; 44 parents/caregivers, 48 children). Wellness Group (n = 92; 47 parents/caregivers, 45 children).
Groups:
- Total: Total of all reporting groups
Arm/Group | NOURISH | Wellness Group | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Continuous [Mean (Standard Deviation); unit: years]
  Adult Age | 38.80 (6.71) | 40.32 (7.81) | 39.90 (7.40)
  Child Age | 8.70 (1.47) | 8.48 (1.53) | 8.60 (1.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 147
  Male | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Child BMI
Description: Children's height and weight were measured and then plotted on the CDC Growth Charts to obtain BMI%ile for age and gender.
Time Frame: Basline, Posttest
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | NOURISH | Wellness Group
Number analyzed (Participants) | 48 | 45
percentile
  Baseline | 98.47 (2.24) | 97.86 (2.67)
  Post-test (12 wks -waves 1-2; 6 weeks-waves 3+) | 98.19 (2.73) | 97.86 (2.61)
Statistical Analysis 1: Comparison: NOURISH vs Wellness Group; Test type: Superiority or Other; p = .008, Chi-squared

2. Secondary Outcome: Child Feeding
Description: The Child Feeding Questionnaire (CFQ) measured parental approaches to and attitudes about feeding their children and the subscale "concern about child's weight" is reported below in the table. The subscale score was calculated by averaging the items (subscale score range: 3 to 15, higher scores represent greater risk). To compare groups, change scores were calculated by subtracting post-test values from baseline values (negative scores indicate decline in parental concern from baseline to post-test).
Time Frame: Basline, Posttest
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOURISH | Wellness Group
Number analyzed (Participants) | 43 | 41
units on a scale | -0.16 (0.44) | -0.03 (0.22)
Statistical Analysis 1: Comparison: NOURISH vs Wellness Group; Test type: Superiority or Other; p = .041, Chi-squared

3. Secondary Outcome: Child Quality of Life
Description: Pediatric Health-Related Quality of Life (PedsQL4.0) change scores from baseline to posttest
  We reported the Total Score. The PedsQL4.0 response scale ranges from 0 - 4. The items are reverse-scored for interpretability and higher scores indicate higher quality of life.
  We used the Total Score, or the mean computed as the sum of all the items over the number of items answered on all the Scales.
  The current report did not provide subscores.
Time Frame: Basline, Posttest
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOURISH | Wellness Group
Number analyzed (Participants) | 48 | 45
units on a scale | 3.47 (12.15) | 1.46 (10.88)
Statistical Analysis 1: Comparison: NOURISH vs Wellness Group; Test type: Superiority or Other; p = .61, Chi-squared

4. Secondary Outcome: Parental BMI
Description: Height and weight were measured by trained staff and used to calculate BMI. Change scores of parental BMI from baseline to posttest were calculated to show difference between treatment arms.
Time Frame: Baseline, Posttest
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | NOURISH | Wellness Group
Number analyzed (Participants) | 44 | 47
kg/m^2 | .42 (1.84) | -.65 (2.96)
Statistical Analysis 1: Comparison: NOURISH vs Wellness Group; Test type: Superiority or Other; p = 0.13, Chi-squared

5. Secondary Outcome: Parental Dietary Intake of Fat
Description: Parents completed a 3 day dietary record which was reviewed by a dietitian and analyzed using the Nutrition Data System Software (NDS-R) to calculate parental fat intake. Change scores were calculated by subtracting post-test values from baseline values; thus, a negative score indicates a greater reduction in fat intake at post-testing.
Time Frame: Baseline, Posttest
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | NOURISH | Wellness Group
Number analyzed (Participants) | 44 | 47
grams | -6.15 (13.66) | -0.42 (15.35)
Statistical Analysis 1: Comparison: NOURISH vs Wellness Group; Test type: Superiority or Other; p = .024, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- NOURISH: The first 2 waves and second 2 waves of participants received a 12 and 6 week face-to-face intervention (NOURISH), respectively. The interventions differed only in duration. They covered the same concepts which are grounded in Social Cognitive Theory (SCT). Throughout the interventions the influence of social learning on behavioral outcomes (e.g., parent's modeling of healthy behavior) was emphasized. Weekly topics provided information about implementing healthy lifestyle behaviors, authoritarian parenting approaches, and strategies for overcoming barriers to change. Parents received pedometers for themselves and 1 of their children. A one-hour booster session was available for all intervention participants 2 months after completion of the interventions.
- Wellness Group: The placebo control group attended a group session moderated by an independent interventionist. This interventionist was blinded to the Specific Aims and hypotheses of this study. The session addressed the role of diet and exercise in pediatric overweight. In addition, parents received pedometers for themselves and 1 of their children. Finally, control participants were mailed publicly available brochures on pediatric overweight on 2 occasions during the study. Control participants were sent home one additional packet of information (essentially a review of previous mail outs) 2 months after post-testing.Followed up for 6 months.
Arm/Group | NOURISH | Wellness Group
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/92
Other Adverse Events (participants affected / at risk) | 0/92 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No